CLINICAL TRIAL: NCT06158165
Title: Evaluating The Cardiovascular Effects of Tourniquet Application
Status: Completed | Type: Observational
Sponsor: Merve Şeker (Other)
Collaborators: Acibadem University (Other)
Responsible Party: Sponsor-Investigator, Merve Şeker, Principal Investigator, Acibadem University
Organization: Acibadem University (Other)
Other Study IDs: AcibademStudy
Record Dates: First submitted 2023-11-18; First posted 2023-12-06 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Orthopedic Disorder; Hemodynamic Instability
Keywords: cardiac cycle efficiency; arterial elastance; dP/dtmax; cardiac power output; tourniquet
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia: Patients undergoing elective unilateral total knee arthroplasty with tourniquet application under the general anesthesia technique
  Interventions: Device: Mostcare (Vytech, Vygon, Padua, Italy)
- Combined Spinal Epidural Anesthesia: Patients undergoing elective unilateral total knee arthroplasty with tourniquet application under the combined spinal epidural anesthesia technique
  Interventions: Device: Mostcare (Vytech, Vygon, Padua, Italy)

INTERVENTIONS:
Device: Mostcare (Vytech, Vygon, Padua, Italy) — Parameters were observed through the utilization of the MostCare (Vytech, Vygon, Padua, Italy) device employing the Pressure Recording Analytic Method (PRAM).

SUMMARY:
The goal of this prospective observational study is to investigate the impact of tourniquet application on cardiac efficiency through the cardiac cycle efficiency parameter and to explore how central regional technique alters this effect compared to general anesthesia.

We aim to answer the following main questions: 1) Does the use of a tourniquet reduce cardiac efficiency? 2) Does the impact of tourniquet use on cardiac efficiency vary with general anesthesia or central regional technique? The patients included in the study will be divided into two groups based on whether they receive general anesthesia or combined spinal epidural anesthesia.The patients' cardiac cycle efficiency and advanced hemodynamic monitoring parameters will be recorded during procedure.

DETAILED DESCRIPTION:
After obtaining ethical committee approval (ATADEK; 2022-14/12), 43 patients undergoing elective unilateral total knee arthroplasty under tourniquet were enrolled in our prospective observational study. Patients were divided into two groups: general anesthesia (Group GA: 22 patients) or combined spinal epidural anesthesia (Group CSEA: 21 patients). Cardiac and vascular parameters were recorded using the new algorithmic application of arterial wave analysis called Pressure Recording Analytical Method (PRAM) at 9 time points: (T1) pre-anesthesia, (T2) post-anesthesia before tourniquet inflation, (T3-8) during tourniquet inflation, and (T9) after tourniquet deflation.

ELIGIBILITY:
Inclusion Criteria:

* Planned for Elective Unilateral Total Knee Arthroplasty Under Tourniquet Application
* Aged 18 and over
* Either general anesthesia (GA) or combined spinal-epidural anesthesia (CSEA) will be administered

Exclusion Criteria:

* Patients under 18 years of age
* Patients with heart failure
* Patients with valve disease
* Patients with rhythm disorders
* Patients with a history of myocardial infarction in the last 3 months
* Patients unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients Scheduled for Elective Unilateral Total Knee Arthroplasty Under Tourniquet Application
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Cardiac Cycle Efficiency (CCE), which measured with the MostCare (Vytech, Vygon, Padua, Italy) device employing the Pressure Recording Analytic Method (PRAM). | 1 minute before and 10 minutes after anesthesia induction, 10-2-30-60 minutes after tourniquet inflation, 1 minute before tourniquet deflation, 1 minute and 5 minutes after tourniquet deflation
  The CCE value must be less than 1. Approaching zero or falling to a negative value indicates a decrease in cardiac efficiency and activation of the myocardial compensation mechanisms. The PRAM minimises artefacts and data variability in patients with haemodynamic instability with its high resolution by acquiring 1000 data per second.
  The CCE parameter, which we utilized to assess the impact of tourniquet application on cardiac efficiency, was measured at the following time points: 1 minute before anesthesia induction (T1), 10 minutes after anesthesia induction, which is 1 minute before tourniquet inflation (T2), 10 minutes after tourniquet inflation (T3), 20 minutes after tourniquet inflation (T4), 30 minutes after tourniquet inflation (T5), 60 minutes after tourniquet inflation (T6), 1 minute before tourniquet deflation (T7), 1 minute after tourniquet deflation (T8), and 5 minutes after tourniquet deflation (T9).

CONTACTS AND LOCATIONS:
Overall Officials: Serap Aktaş yıldırım, doctor, Study Chair — Acibadem University; Bülent Güçyetmez, doctor, Study Chair — Acibadem University; Halim Ulugöl, doctor, Study Chair — Acibadem University; Fevzi Toraman, doctor, Study Chair — Acibadem University
Locations (1):
- Acibadem University, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The Informed Consent Form will be shared
Supporting Information: ICF
Time Frame: September 2022 and April 2023
Access Criteria: If requested, the Informed Consent Form will be shared via email